CLINICAL TRIAL: NCT07253818
Title: Transthoracic Echocardiography as the Reference for Validating Non-invasive Hemodynamic Monitoring During Passive Leg Raising in Term Pregnancy
Brief Title: Passive Leg Raising in Term Pregnancy on Hemodynamic Monitoring - Validating With Transthoracic ECHO (LG-ECHO)
Acronym: (LG-ECHO)
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawned because of lack of relevant devices in the study center
Sponsor: Ayse Zeynep Turan Civraz (Other Government)
Responsible Party: Sponsor-Investigator, Ayse Zeynep Turan Civraz, Assoc. Prof. Dr., Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Other Study IDs: AS-01-OBS
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Maternity; Pregnancy; Labor and Delivery; Hemodynamic Changes
Keywords: hemodynamic changes; pregnancy; clearsight; transthoracic echocardiography; Passive Leg Raising Maneuver
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: ClearSight™ System — ClearSight™ is FDA 510(k) cleared for non-invasive measurement of blood pressure and derived hemodynamic parameters in adults (≥18 years) and pediatric patients ≥12 years when used with EV1000 or HemoSphere Baseline, during passive leg raising (PLR) and after PLR measurements will be acquired. Data will be continuously recorded for 5 minutes at 60-second intervals using a dedicated monitor (EV1000™).
Device: Transthoracic Echocardiography — This study uses transthoracic echocardiography (TTE), which is a non-invasive imaging modality All measurements will be obtained with participants in the 15° left tilt position in order to minimize inferior vena cava compression from the gravid uterus and to avoid haemodynamic fluctuations associated with positional changes Initially, the left ventricular outflow tract (LVOT) diameter will be obtained at end-expiration in the parasternal long-axis view, measured from the inner edge to inner edge of the aortic annulus. Subsequently, the LVOT velocity-time integral (LVOT-VTI) will be assessed using pulsed-wave Doppler, with the sampling volume positioned at the centre of the LVOT in the apical five-chamber view. LVOT diameter will be measured from the parasternal long-axis view (inner-edge to inner-edge, mid-systole), with the average of two measurements recorded.
  Measurements will be recorded at three timepoints: baseline at the end of PLR, after PLR
Procedure: Passive Leg Raising (PLR) Maneuver — This manoeuvre acts as a rapid, transient, and reversible "auto-fluid challenge" by mobilizing blood from the venous reservoir of the lower extremities into the central circulation. The resulting temporary increase in preload can augment cardiac output in preload-responsive patients through the Frank-Starling mechanism .
  An electronically adjustable bed, capable of altering position without requiring active movement from the participant, will be utilized in the study. Baseline hemodynamic recordings will be taken following 5 minutes of rest in supine position with 15° left tilt, and the head of the bed elevated to 45°. Subsequently, the head section of the bed will be swiftly returned to a flat position, while the leg section will be elevated to 45°, thereby achieving passive leg raising. Hemodynamic variables will be measured around 90 seconds after PLR will be compared with baseline values.

SUMMARY:
This prospective observational validation study aims to evaluate the agreement and diagnostic accuracy of ClearSight™ compared with transthoracic echocardiography (TTE) during PLR in term pregnant women.

The ultimate goal is to determine whether ClearSight™ can reliably identify preload responsiveness in term pregnant women compared with the echocardiographic gold standard. The clinical implication is that, if validated, ClearSight™ may reduce unnecessary or harmful fluid administration by accurately detecting preload reserve, and improve maternal safety in peripartum care by providing obstetric anesthesiologists with reliable bedside monitoring tools.

DETAILED DESCRIPTION:
Background Pregnancy is characterized by profound hemodynamic changes, which complicate perioperative monitoring and fluid therapy. Non-invasive cardiac output monitoring device, ClearSight™ system, provides continuous stroke volume estimates, but their reliability in pregnant women remains uncertain. Passive leg raising (PLR) is a reversible preload test that can elucidate fluid responsiveness without fluid administration. To date, no study has simultaneously validated ClearSight™ against echocardiographic reference standards during PLR in term pregnant women.

Methods This is a prospective, single-centre, method-comparison and diagnostic accuracy study in term pregnant women (≥37 weeks). Simultaneous ClearSight™ and transthoracic echocardiography (TTE) measurements will be obtained at baseline, during PLR, and during recovery. The primary outcome is agreement between ClearSight™-derived stroke volume index (SVI) changes and TTE-derived Left Ventricular Outflow Tract - Velocity Time Integral (LVOT-VTI) changes during PLR. Secondary outcomes include trending ability and diagnostic accuracy of ClearSight™ Δ%SVI for detecting PLR responders. Four-quadrant and polar plot analyses are the parameters for advanced hemodynamic monitoring methods used in echocardiography to assess fluid responsiveness and cardiac output (CO) trending Sample size: 60 participants, providing at least 180 paired observations.

Conclusions This study will establish whether ClearSight™ can reliably detect preload responsiveness in term pregnant women. Findings could support safer, real-time, non-invasive hemodynamic management during obstetric anaesthesia and maternal critical care.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnant patients
* Singleton pregnancy at ≥37+0 weeks of gestation.
* Maternal age between 18 and 45 years.
* Hemodynamically stable and in sinus rhythm.
* Ability to provide verbal and written informed consent.

Exclusion Criteria:

* Hypertensive disorders of pregnancy, significant valvular or congenital heart disease, cardiomyopathy, or persistent arrhythmias.
* Multiple gestation (i.e., Twin pregnancy and above)
* Endocrine or hematologic conditions likely to affect hemodynamics, including diabetes with or without autonomic neuropathy, thyroid storm, or severe anemia (hemoglobin <8 g/dL).
* Active labor with pain or current infusion of uterotonic or vasoactive agents.
* Ruptured membranes with frequent contractions or indications for emergent delivery.
* Inadequate transthoracic echocardiographic imaging windows at screening.
* Emergency or STAT (statim) Cesarean Deliveries

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study will be conducted on pregnant women
Study Population: Patients will be enrolled when they come to the OB clinic for evaluation and the consents will be obtained. Patients are instructed during consent to abstain from caffeine/nicotine (≥4h) and heavy meals (≥6h). This is feasible as women are already required to fast preoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Agreement between ClearSight™-derived stroke volume index (SVI) changes and TTE-derived Left Ventricular Outflow Tract - Velocity Time Integral (LVOT-VTI) changes during PLR. | During PLR
  The primary outcome is agreement between ClearSight™-derived stroke volume index (SVI) changes and TTE-derived Left Ventricular Outflow Tract - Velocity Time Integral (LVOT-VTI) changes during PLR.

SECONDARY OUTCOMES:
Trending ability and diagnostic accuracy of ClearSight™ Δ%SVI for detecting PLR responders | During PLR
  Trending ability and diagnostic accuracy of ClearSight™ Δ%SVI for detecting PLR responders

CONTACTS AND LOCATIONS:
Overall Officials: Ayten Saracoglu, Prof. MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville (Shands Hospital), Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vartun A, Flo K, Acharya G. Effect of passive leg raising on systemic hemodynamics of pregnant women: a dynamic assessment of maternal cardiovascular function at 22-24 weeks of gestation. PLoS One. 2014 Apr 14;9(4):e94629. doi: 10.1371/journal.pone.0094629. eCollection 2014. PMID 24732308
- [Background] Quinones MA, Otto CM, Stoddard M, Waggoner A, Zoghbi WA; Doppler Quantification Task Force of the Nomenclature and Standards Committee of the American Society of Echocardiography. Recommendations for quantification of Doppler echocardiography: a report from the Doppler Quantification Task Force of the Nomenclature and Standards Committee of the American Society of Echocardiography. J Am Soc Echocardiogr. 2002 Feb;15(2):167-84. doi: 10.1067/mje.2002.120202. No abstract available. PMID 11836492
- [Background] Duclos G, Granier S, Hili A, Blanc J, Einav S, Leone M, Zieleskiewicz L. Performance of non-invasive stroke volume variation during passive leg raising as a predictor of hypotension following induction of spinal anesthesia for elective cesarean delivery: a single cohort study. Int J Obstet Anesth. 2022 May;50:103251. doi: 10.1016/j.ijoa.2021.103251. Epub 2021 Dec 30. PMID 35074676
- [Background] Duclos G, Hili A, Resseguier N, Kelway C, Haddam M, Bourgoin A, Carcopino X, Zieleskiewicz L, Leone M. Clearsight use for haemodynamic monitoring during the third trimester of pregnancy - a validation study. Int J Obstet Anesth. 2018 Nov;36:85-95. doi: 10.1016/j.ijoa.2018.04.009. Epub 2018 May 8. PMID 30392653
- [Background] Marques NR, Martinello C, Kramer GC, Costantine MM, Vadhera RB, Saade GR, Hankins GD, Pacheco LD. Passive leg raising during pregnancy. Am J Perinatol. 2015 Mar;32(4):393-8. doi: 10.1055/s-0034-1389089. Epub 2014 Sep 21. PMID 25241109
- [Background] Herrera S, Kuhlmann-Capek MJ, Rogan SC, Saad AF, Saade GR, Hankins GDV, Pacheco LD. Stroke Volume Recruitability during the Third Trimester of Pregnancy. Am J Perinatol. 2018 Jul;35(8):737-740. doi: 10.1055/s-0037-1615788. Epub 2017 Dec 26. PMID 29278864
- [Background] Vartun A, Flo K, Wilsgaard T, Acharya G. Maternal functional hemodynamics in the second half of pregnancy: a longitudinal study. PLoS One. 2015 Aug 10;10(8):e0135300. doi: 10.1371/journal.pone.0135300. eCollection 2015. PMID 26258418
- [Background] Monnet X, Teboul JL. Prediction of fluid responsiveness in spontaneously breathing patients. Ann Transl Med. 2020 Jun;8(12):790. doi: 10.21037/atm-2020-hdm-18. PMID 32647715
- [Background] Helmer P, Helf D, Sammeth M, Winkler B, Hottenrott S, Meybohm P, Kranke P. The Use of Non-Invasive Continuous Blood Pressure Measuring (ClearSight(R)) during Central Neuraxial Anaesthesia for Caesarean Section-A Retrospective Validation Study. J Clin Med. 2022 Aug 2;11(15):4498. doi: 10.3390/jcm11154498. PMID 35956113
- [Background] Akkermans J, Diepeveen M, Ganzevoort W, van Montfrans GA, Westerhof BE, Wolf H. Continuous non-invasive blood pressure monitoring, a validation study of Nexfin in a pregnant population. Hypertens Pregnancy. 2009 May;28(2):230-42. doi: 10.1080/10641950802601260. PMID 19437233
- [Background] Lihme F, Basit S, Persson LG, Larsen MO, Lauridsen KH, Lykke JA, Andersen AS, Halse K, Thorsen-Meyer A, Melbye M, Wohlfahrt J, Boyd HA. Reference ranges for third-trimester maternal cardiovascular function parameters measured in normotensive pregnant women using a non-invasive cardiac output monitor: A study based on data from the prospective PEACH cohort study. BJOG. 2024 Mar;131(4):463-471. doi: 10.1111/1471-0528.17667. Epub 2023 Sep 21. PMID 37735094
- [Background] McLaughlin K, Wright SP, Kingdom JCP, Parker JD. Clinical Validation of Non-Invasive Cardiac Output Monitoring in Healthy Pregnant Women. J Obstet Gynaecol Can. 2017 Nov;39(11):1008-1014. doi: 10.1016/j.jogc.2017.02.015. Epub 2017 Jul 18. PMID 28733057
- [Background] Ling HZ, Gallardo-Arozena M, Company-Calabuig AM, Nicolaides KH, Kametas NA. Clinical validation of bioreactance for the measurement of cardiac output in pregnancy. Anaesthesia. 2020 Oct;75(10):1307-1313. doi: 10.1111/anae.15110. Epub 2020 May 29. PMID 32469423
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Cornette J, Laker S, Jeffery B, Lombaard H, Alberts A, Rizopoulos D, Roos-Hesselink JW, Pattinson RC. Validation of maternal cardiac output assessed by transthoracic echocardiography against pulmonary artery catheterization in severely ill pregnant women: prospective comparative study and systematic review. Ultrasound Obstet Gynecol. 2017 Jan;49(1):25-31. doi: 10.1002/uog.16015. Epub 2016 Nov 28. PMID 27404397
- [Background] Bijl RC, Valensise H, Novelli GP, Vasapollo B, Wilkinson I, Thilaganathan B, Stohr EJ, Lees C, van der Marel CD, Cornette JMJ; International Working Group on Maternal Hemodynamics. Methods and considerations concerning cardiac output measurement in pregnant women: recommendations of the International Working Group on Maternal Hemodynamics. Ultrasound Obstet Gynecol. 2019 Jul;54(1):35-50. doi: 10.1002/uog.20231. PMID 30737852